CLINICAL TRIAL: NCT02197455
Title: Tofacitnib for the Treatment of Alopecia Areata and Variants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1407014260
Record Dates: First submitted 2014-07-18; First posted 2014-07-22 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Alopecia Areata (AA); Alopecia Totalis (AT); Alopecia Universalis (AU)
MeSH Terms: conditions — Alopecia Areata; Alopecia universalis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tofacitinib Administration (Experimental): 5 mg of Tofacitinib will be taken by mouth twice daily for 3 months.
  Interventions: Drug: Tofacitinib Administration

INTERVENTIONS:
Drug: Tofacitinib Administration — 5 mg of Tofacitinib will be taken by mouth twice daily for 3 months.

SUMMARY:
The purpose of this study is to investigate the ability of tofacitinib citrate, a Janus kinase inhibitor, to generate hair regrowth in patients with moderate to severe alopecia areata and its variants.

DETAILED DESCRIPTION:
This study is an open-label pilot study. Participants will be treated with oral tofacitinib for a maximum of 5 months. Participants will be evaluated at 3 months after completion of therapy to evaluate for durability of response, late response and/or late adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Diagnosis of alopecia areata with >50% scalp involvement, alopecia totalis, or alopecia universalis
* Hair loss present for at least 6 months
* No treatment for alopecia areata in past 2 months
* No evidence of hair regrowth
* Females of childbearing potential must use birth control while taking the medication and there must be a negative pregnancy test documented prior to starting the medication

Exclusion Criteria:

* Age <18 years old
* Patients have received treatment known to affect alopecia areata within 2 months of enrolling in the study
* Patients with a history of malignancy (except history of successfully treated basal cell or squamous cell carcinoma of the skin)
* Patients known to be HIV or hepatitis B or C positive
* Patients with positive tuberculin skin test or positive QuantiFERON TB test
* Patients with leukopenia or anemia
* Patients with renal or hepatic impairment
* Patients with peptic ulcer disease
* Patients taking immunosuppressive medications, including but not limited to prednisone, methotrexate, mycophenolate mofetil, azathioprine, tacrolimus, cyclosporine, or TNH-alpha inhibitors
* Women of childbearing potential who are unable or unwilling to use birth control while taking the medication
* Women who are pregnant or nursing

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett King, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kennedy Crispin M, Ko JM, Craiglow BG, Li S, Shankar G, Urban JR, Chen JC, Cerise JE, Jabbari A, Winge MC, Marinkovich MP, Christiano AM, Oro AE, King BA. Safety and efficacy of the JAK inhibitor tofacitinib citrate in patients with alopecia areata. JCI Insight. 2016 Sep 22;1(15):e89776. doi: 10.1172/jci.insight.89776. PMID 27699252

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tofacitinib Administration
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tofacitinib Administration
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (15.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Severity of Alopecia Tool (SALT) Score
Description: SALT score range is from 0 (no hair loss) to 100 (100% hair loss)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percent change in SALT score
Arm/Group | Tofacitinib Administration
Number analyzed (Participants) | 30
percent change in SALT score | 22.8 (30.3)

2. Secondary Outcome: Mean Change in Skindex 16 Scores
Description: Skindex 16 is a quality of life questionaire with a range of 0-100 wherein 1 is not bothered by the condition and 100 is always bothered by the condition
Time Frame: 3 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Tofacitinib Administration
Number analyzed (Participants) | 30
units on a scale | -20.3 [-61.6 to 7.3]

ADVERSE EVENTS:
Arm/Group | Tofacitinib Administration
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 18/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib Administration (N=30)
cold (Infections and infestations) | 3
sinus infection (Infections and infestations) | 2
headache (Nervous system disorders) | 3
abdominal pain (Gastrointestinal disorders) | 2
acne (Skin and subcutaneous tissue disorders) | 4
fatigue (General disorders) | 2
night sweats (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No